CLINICAL TRIAL: NCT06378515
Title: Physical Activity, Sleep and Brain Health Based on the Glymphatic System
Status: Recruiting | Type: Observational
Sponsor: University of Valencia (Other)
Collaborators: University of Oulu (Other)
Responsible Party: Principal Investigator, Raquel Faubel Cava, Lecturer in Physiotherapy, University of Valencia
Other Study IDs: Glymphactive
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Brain Diseases
Keywords: glympathic system; brain health; physical activity; neurohydrodynamics
MeSH Terms: conditions — Brain Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Physical activity, postural changes and cognitive tasks — 1. Measuring while patients are sitting in rest for 5 minutes.
  2. Supine to stand test: lying down (5 min) standing up (5 min)
  3. Repeated sit stand test: sitting (10 sec) ↔ standing (10 sec), changing position every 10 seconds for 5 minutes.
  4. Paced breathing in sitting position: letting patients breath 6 breaths/minute (0.1Hz) for 5 minutes.
  5. Breath hold manoeuvre in sitting position: 60s normal breathing, then 32s breath hold + 88s normal breathing repeated 3 times.
  6. Arithmetic stress test by giving the subject single digit addition. To give the pressure, subject needs to do as many as possible calculation within 1 minute with 1 minute break. This is repeated 3 times.

SUMMARY:
This study is aiming to analyze the impact of physical activity on neurohydrodynamics and glymphatic activity on young adults. This study is designed as a multicenter descriptive observational study with information collection at two different times: before performing a short exercise routine and during its performance using a wearable wireless device Glymphometer.

DETAILED DESCRIPTION:
The glymphatic system was discovered in 2013 as a brain mechanism for the elimination of protein waste in the central nervous system. Scientific findings indicate that an abnormality in this system involves a slow accumulation of protein waste, neurological inflammation, leaks in the blood-brain barrier, and finally neuronal degeneration due to the progressive loss of neurons in the central nervous system. Brain fluid dynamics, particularly those related to cerebrospinal fluid, have been shown to play an important role in brain health and the progression of neurodegenerative diseases. The Glymphometer is a device that allows the evaluation of brain health in a novel way, as it allows the monitoring of brain fluid dynamics and could allow early detection of abnormalities in the glymphatic system. This technology makes it easy to monitor brain health and allows you to set actions for a healthier lifestyle. It also makes it possible to monitor the effectiveness of emerging therapies to avoid or reduce the risk of neurological diseases. In the long term, this could allow for more cost-effective prevention tools. This device has been used in numerous research projects and is also closely related to other projects funded by the European Commission currently underway such as Neurodegenerative Disease Research (JPND). The data generated by these wearable devices will also be useful for healthcare systems as such data can be collected in other situations such as during sleep, exercise or at work. These devices will be used both at the diagnostic level and also to monitor the impact of neurological therapies, allowing for more personalized treatments. The Glymphometer has previously been used in studies that have looked at the impact of stress on brain health. Physical activity and exercise are other lifestyle factors that have an influence on brain health, as shown by preclinical studies and recent reviews on the glymphatic system, and have been proposed as preventive therapy and treatment for dementia due to their impact on the glymphatic system. The existing literature shows that lifestyle factors such as sleep, physical activity or stress can be highly relevant to brain health, but there is not enough scientific evidence based on continuous measurements of how they affect it.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in a bachelor's degree from one of the universities participating in the study.
* Students who consent to participate in the study indicating that they have been informed of all relevant aspects of the study.

Exclusion Criteria:

* Students under the age of 18.
* Students with cognitive or sensory difficulties or with insufficient command of the language that, in the opinion of the recruiting professional, makes it difficult to understand the questions raised in the surveys, scales or instruments used in the study.
* Who are participating at the time of recruitment in a clinical trial or experimental study. Participation in observational studies will not be an exclusion criterion

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity.
Study Population: University students
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Brain health | Basal, during 15 minutes
  The data collected through the Glymphometer allows us to obtain the variable known as the G-index, which describes the activity of the glymphatic system. This G-index is based on 14 (patented) algorithms. The G-index ranges from 0 to 100, with higher brain health the higher the score
  Brain health through the G-Index. Data collected through the Glymphometer allows us to obtain the variable known as the G-index, which describes the activity of the glymphatic system. This G-index is based on 14 (patented) algorithms and ranges from 0 to 100, with higher brain health the higher the score.

SECONDARY OUTCOMES:
Physical activity (habitual) | Basal
  Physical activity developed during the last 7 days using the short version of validated questionnaire IPAQ (International Physical Activity Questionnaire)
Sleep duration | Basal
  Number of hours of sleep habitual (including naps) specifically in weekdays and weekends. Collected by indirect methods using self-reported questions.
Sleep Quality | Basal
  Brief Version of the Pittsburgh Sleep Quality Index (B-PSQI)
Chronotype | basal
  Morning or night preferences collected by the short version of validated questionnaire MEQ (rMEQ)
Self-reported health status | Basal
  Self-reported by the participant using a specific question about their health status during the last 12 months
Other variables | Basal
  Other variables of interest collected reported by the participant through an ad hoc questionnaire: height and weight, age, sex, chronic conditions diagnosed, country of residence, academic degree studied, years at university, tobacco and alcohol consumption, cohabitation (alone, in family, shared), complementary activities (hours per week dedicated to other activities outside the university in the last month such as work, Other regulated studies, volunteering, family care...

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Faubel, PhD, Principal Investigator — Universitat de València
Locations (1):
- Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data of the participants is planned to be shared with other researchers for scientific reasons.
Supporting Information: Study Protocol, CSR
Time Frame: after the data collection
Access Criteria: Data will be available based on the criteria of the main researcher